CLINICAL TRIAL: NCT04663659
Title: The Effect of Diabetes Mellitus on Mortality in Patients Hospitalized in the COVID Intensive Care Unit in the COVID-19 Pandemic
Brief Title: The Effect of Diabetes Mellitus on Mortality of Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nermin Balta Başı, medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 1559
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Diabetes Mellitus
MeSH Terms: conditions — COVID-19; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic group: Patients over the age of 18 with diabetes mellitus in intensive care unit
  Interventions: Other: no intervention
- non-diabetic group: Patients over the age of 18 without diabetes mellitus in intensive care unit
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The study includes patients over 18 years old who were hospitalized in our covid intensive care unit between March 16 and May 16, 2020.

Retrospective records were examined by examining the electronic data files of the patients.

Polymerase Chain Reaction (PCR) tests performed with nasopharyngeal swab taken from the person, which is the standard diagnostic method, and also the diagnosis of infection symptoms, risk factors and thoracic CT scans indicating pneumonia were diagnosed.

Patients over 18 years of age with and without a medical history of DM in their history were identified and compared in 2 groups.

DETAILED DESCRIPTION:
The study includes patients over 18 years old who were hospitalized in our covid intensive care unit between March 16 and May 16, 2020.

Retrospective records will be examined by examining the electronic data files of the patients.

Polymerase Chain Reaction (PCR) tests performed with nasopharyngeal swab taken from the person, which is the standard diagnostic method, and also the diagnosis of infection symptoms, risk factors and thoracic CT scans indicating pneumonia were diagnosed.

Patients over 18 years of age with and without a medical history of DM in their history will be identified and compared in 2 groups.

Demographic data such as age, gender, Body Mass Index (BMI) of all patients, presence of additional comorbid disease, blood glucose values during hospitalization in intensive care, ferritin, C-Reactive Protein (CRP), respiratory support methods (nasal oxygen, nasal high flow, non-invasive mechanical ventilation, intubation), length of stay in intensive care unit, and mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age

Exclusion Criteria:

* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with and without a medical history of DM in their history will be identified and compared in 2 groups
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Mortality | 3 months
  Mortality rates of patients
length of stay in intensive care | 3 months
  The time between admission to intensive care unit and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nermin Balta Basi, Principal Investigator — Sisli Hamidiye Etfal Education and Training Hospital
Locations (1):
- SisliHamidiye Etfal Education and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided